CLINICAL TRIAL: NCT02594995
Title: The Impact of NBP on the Collateral Circulation in Acute Acute Internal Carotid Artery(ICA)/Middle Cerebral Artery(M1) Occlusion
Brief Title: The Impact of NBP on the Collateral Circulation in ICA/M1 Occlusion
Acronym: INCIMO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SAHZJUNeuro
Record Dates: First submitted 2015-10-22; First posted 2015-11-03 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2016-04

CONDITIONS: Cerebrovascular Occlusion; Collateral Blood Circulation; Anterior Cerebral Circulation Infarction
MeSH Terms: conditions — Cerebrovascular Disorders; Brain Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- NBP in thrombolysis group (Experimental): NBP 25mg bid for 2 weeks administered after 24 hours after receiving recombinant plasminogenactivator(rt-PA) thrombolysis
  Interventions: Drug: NBP
- NBP group (Experimental): NBP 25mg bid for 2 weeks administered for the patients who do not receive rt-PA
  Interventions: Drug: NBP
- Control group (No Intervention): Control group not receiving rt-PA thrombolysis, receiving basic therapy for acute stroke, e.g. aspirin/clopidogrel and lipid-lowering therapy
- Control in thrombolysis group (No Intervention): Control group receiving rt-PA thrombolysis

INTERVENTIONS:
Drug: NBP
  Arms: NBP group; NBP in thrombolysis group

SUMMARY:
Stroke is the first leading cause of death in China, and is responsible for almost 22.4% of deaths. In approximately 80% of cases stroke is ischaemic, i.e. caused by disruption of blood flow to part of the brain from an acute arterial occlusion. Survival of penumbral tissue distal to an arterial occlusion depends on collateral circulation via the Circle of Willis and leptomeningeal anastomises. Collateral flow is dynamic and failure is associated with infarct growth. The presence of adequate collaterals has been shown to be associated with age, history of statin use, and non-hypertension. Dl-3-n-butylphthalide (NBP), isolated from the seeds of celery, and found to exert protective effects against ischemic brain and increase leptomeningeal blood flow. This study investigate whether NBP injection prescribed during acute stroke will have a significant effect to improve collateral circulation in patients of anterior circulation occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥ 18 years old;
2. Acute occlusion of M1 or intracranial internal carotid artery within 72 hours;
3. For patients who receive recombinant tissue-type plasminogenactivator therapy, the arterial occlusive lesion scale of 24-72 hours post-thrombolysis imaging should be 0 or 1;
4. Ischemic stroke with National Institutes of Health Stroke Scale ≥ 4;
5. Baseline mRS before this stroke onset less than 2;
6. Able and willing to comply with study requirements;
7. Signed informed consent by patients self or legally authorized representatives.

Exclusion Criteria:

1. Cerebral hemorrhage;
2. Posterior circulation infarction;
3. Severe tendency of hemorrhage, such as thrombocytopenia, leukemia, allergic purpura;
4. Currently using urinary kallidinogenase or alprostadil;
5. Be allergic to NBP or celery;
6. Impaired liver function (alanine aminotransferase or glutamic oxalacetic transaminase ≥ 3×upper limit of normal) or renal function (serum creatinie ≥ 1.5mg/dl);
7. Patients with evidence of severe congestive heart failure or history of end-stage cardiovascular disease (e.g. congestive heart failure New York Heart Association Class III or IV);
8. Metastatic neoplasm or multiple organ failure;
9. Pregnancy or breastfeeding;
10. History of mental instability or dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2015-07; Primary Completion 2016-09-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
the percentage of patients with modified Rankin Score (mRS) equivalent to or less than 2 | 3 months

SECONDARY OUTCOMES:
rLMC scale of Collateral circulation | 2 weeks, 3 months
  We use regional leptomeningeal score(rLMC) score to measure collateral circulation.rLMC score is based on scoring pial and lenticulostriate arteries in 6 ASPECTS regions(M1-6) plus anterior cerebral artery region and basal ganglia. Pial arteries in the Sylvian sulcus are scored 0,2, or 4.
NIHSS score | 1 week, 2 weeks, 3 months
Hemorrhageic complications including intracranial, digestive tract | 2 weeks, 3 months
New stroke or transient ischemic attack(TIA) | 3 months
complete blood count | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Min Lou, Ph.D, M.D., Study Chair — second affiliated hospital of Zhejiang University, school of medicine
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China